CLINICAL TRIAL: NCT02333695
Title: Medical Device for Magnetic Therapy for Spinal Cord Injuries (SCIMAG)
Brief Title: Medical Device for Magnetic Therapy for Spinal Cord Injuries (SCI)
Acronym: SCIMAG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: American Society Of Thermalism And Climatology Inc (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Gavionerrvemag
Record Dates: First submitted 2015-01-05; First posted 2015-01-07 (Estimated); Last update posted 2015-01-07 (Estimated); Status verified 2015-01

CONDITIONS: Spinal Cord Injury; Stroke
Keywords: SCI, Spinal Cord Injury, Stroke
MeSH Terms: conditions — Spinal Cord Injuries; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Spinal Magnetic Stimulation (Experimental): Spinal Magnetic Stimulation (SMS) is a relatively new way to use magnetism to affect the spinal cord. It is non-invasive, meaning that the procedure does not require any type of surgery; rather, it is conducted by transmitting magnetic pulses through the Spinal Cord by pressing a machine against the back.
  Interventions: Device: Spinal Magnetic Stimulation

INTERVENTIONS:
Device: Spinal Magnetic Stimulation — Spinal Magnetic Stimulation (SMS) is a relatively new way to use magnetism to affect the spinal cord. It is non-invasive, meaning that the procedure does not require any type of surgery; rather, it is conducted by transmitting magnetic pulses through the Spinal Cord by pressing a machine against the back.
  Other Names: SMS

SUMMARY:
A medical device for magnetic therapy for spinal cord injuries (SCI) will be disclosed. The apparatus comprises a combination of several magnets enclosed in a supportive cover. The magnets are placed in a proper position and their polarity can be changed at any time without any difficulty.

DETAILED DESCRIPTION:
A medical device for magnetic therapy for spinal cord injuries (SCI) will be disclosed. The apparatus comprises a combination of several magnets enclosed in a supportive cover. The magnets are placed in a proper position and their polarity can be changed at any time without any difficulty.

The device provides a source of stimulation for the nerve to achieve therapeutic results and rehabilitation of patients with spinal trauma or stroke.

A spinal cord injury - damage to any part of the spinal cord or nerves at the end of the spinal canal - often causes permanent changes in strength, sensation and other body functions below the site of the injury.

Many scientists are optimistic that advances in research will someday make the repair of spinal cord injuries possible. Research studies are ongoing around the world. In the meantime, treatments and rehabilitation allow many people with a spinal cord injury to lead productive, independent lives.

The effects of SCI depend on the type of injury and the level of the injury. SCI can be divided into two types of injury - complete and incomplete.

Complete: A complete injury means that there is no function below the level of the injury; no sensation and no voluntary movement. Both sides of the body are equally affected.

Incomplete: An incomplete injury means that there is some functioning below the primary level of the injury. A person with an incomplete injury may be able to move one limb more than another, may be able to feel parts of the body that cannot be moved, or may have more functioning on one side of the body than the other. With the advances in acute treatment of SCI, incomplete injuries are becoming more common.

Spinal Magnetic Stimulation (SMS) is a relatively new way to use magnetism to affect the spinal cord. It is non-invasive, meaning that the procedure does not require any type of surgery; rather, it is conducted by transmitting magnetic pulses through the Spinal Cord by pressing a machine against the back.

The Long term goal of this research project is the implementation of an effective, inexpensive therapy in patients with spinal cord injury. Another objective is the development of a cheap, presentable and comfortable magnetic device that causes neural stimulation to stop and reversing the signs and symptoms of Spinal Cord injury.

The short-term objective is to prove that magneto stimulation is an intervention that reverses the signs and symptoms of Spinal Cord injury in an early and moderate State

ELIGIBILITY:
Inclusion Criteria:

* informed consent;
* persons with confirmed and verified lesion of the central nervous system

Exclusion Criteria:

* Identification of the study a total intolerance to a pulsed magnetic field;
* Development after inclusion of acute myocardial infarction and acute ischemic;
* Installation of the pacemaker, intracardiac catheters or operations on the brain, requiring the abandonment of metal objects in the cranial cavity;
* Pregnancy;
* Enhancement of the patient, which requires the maintenance of vital functions by hardware (mechanical ventilation, continuous application infusomats);
* The emergence of an epileptic seizure ;
* Failure of the patient to continue participation in the study;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-01; Primary Completion 2015-08 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Reduction Hiperrelexia | 30 days

SECONDARY OUTCOMES:
Stimulate an erection | 45 days
Stimulate bowel movements | 30 days
Stimulate bladder emptying | 30 days

OTHER OUTCOMES:
Reduce muscle spasticity following upper motor neuron lesions | 45 days
Induce cough to prevent respirator infections. | 45 days

CONTACTS AND LOCATIONS:
Overall Officials: Garis Silega, MD, Principal Investigator — America Society of thermalism
Locations (1):
- Gaviota Clinic, Newark, New Jersey, United States